CLINICAL TRIAL: NCT01359215
Title: Is Pediatric Anesthesia Associated With Long-term Hippocampal Dysfunction?
Brief Title: Childhood Anesthesia and Cognitive Function
Acronym: UCSF-Anes-01
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01926
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Cognitive Deficits; Cognitive Ability, General
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Children who received an anesthetic prior to age 2
- Control: Children who have never been anesthetized

SUMMARY:
The purpose of this study is to determine whether pediatric anesthesia is associated with long-term hippocampal dysfunction

DETAILED DESCRIPTION:
Contrary to a longstanding belief, anesthesia has lasting effects on the neonatal brain. In rats anesthesia causes death of brain cells, ill-timed conversion of stem cells to nerve cells and a certain kind of brain defect up to 8 months later. This brain defect is called a hippocampal deficit because it resembles the type of defect that people have when a structure in the brain called the hippocampus has been injured, removed or is no longer functioning. However, to date it is unknown if anesthesia given to human infants causes a lasting hippocampal deficit, which might manifest itself as memory problems and academic failure despite normal intelligence. The investigators will test the hypothesis that anesthesia for more than 2h given to children of less than 2 years of age without coexisting diseases of the brain or the heart causes long-term impairment of hippocampal function. Using state of the art hippocampal and general brain function testing the investigators will compare hippocampal dependent and hippocampal independent memory as well as general cognitive function and emotional state in 10 year-old children that underwent at least a 2h anesthetic at less than 2 years with that of a matched control group that did not undergo an anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia at less than 2 years of age
* Anesthetic time greater than 2 hours
* ASA I or II
* Induction with Propofol or Sevoflurane +/- N2O
* Maintenance with a volatile agent (sevoflurane, isoflurane, desflurane) +/- N2O

Exclusion Criteria:

* Neurosurgery
* Known genetic syndrome
* Any other anesthetic agents (ketamine, meperidine, barbiturates, etomidate, methoxyflurane, methadone, lorazepam)
* Low birthweight (<25%ile)
* Gestational age , 36 weeks
* color blindness
* h/o CNS disease
* cancer
* head trauma
* congenital heart disease
* ASA III or IV
* intra-operative hypotension (<30% baseline for > 5 min)
* Bradycardia (<30% baseline for > 5 min)
* Hypoxemia (Blood Oxygen Saturation <93% for > 5 min)
* Hypercarbia (pCO2 > 60 mm Hg > 5 min)
* Dysthermia (deviation from 36.5 deg C by > 1.5 deg C at any time)
* Puberty

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who received an anesthetic early in life
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Recollection | 6-12 years of age
  Subjects who received and anesthetic during the first two years of life and controls are given a cognitive test at 6 to 12 years of age

SECONDARY OUTCOMES:
Familiarity, Child behavioral checklist | 6-12 years of age
  cognitive testing

CONTACTS AND LOCATIONS:
Overall Officials: Greg Stratmann, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of Califoria, Davis, Davis, California
  - Univeristy of California, San Francisco, San Francisco, California